CLINICAL TRIAL: NCT04799366
Title: Contractile Properties of Hypertrofic Muscles in Patients With Non-Dystrophic Myotonia
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Laura Nørager Jacobsen, BSc, Rigshospitalet, Denmark
Other Study IDs: H-18023049-1
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Non-Dystrophic Myotonia; Myotonia Congenita
MeSH Terms: conditions — Myotonia Congenita

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MC: MC patients with either dominant (Thomsens) or recessive (Becker) myotonia.
- Healthy Controls: Healthy controls age- and gender matched.

SUMMARY:
In myotonia congenita (MC), mutations in the CLCN1 gene coding a key chloride channel expressed in muscle cells cause myotonia. On examination, the myotonia can be demonstrated as delayed muscle relaxation of muscle contractions after mechanical stimulations. Existing literature describe no muscle weakness in MC patients, however a recent muscle MRI study in non-dystrophic myotonia patients found structural abnormalities in affected muscles when examined using T1 and STIR imaging. The question remains whether the signs of structural changes in the muscle are merely due to the myotonia, or long-term effects of elevated stress of the tissue, and if so, whether those changes lead to clinically significant loss of contractile properties of the muscle.

This study examines if the contractile properties of myotonic muscles are impaired in MC patients. 40 patients with Thomsens disease (n=20) and Beckers disease (n=20), respectively, will be included along with 20 healthy controls. Peak muscle torque is measured in the hand by hand dynamometer and in the thigh and calf muscles with a Biodex System 4 Pro Dynamometer and the cross-sectional area of the muscles are examined on T1-weighed and Dixon-MRI-scan. With the obtained data peak torque in strength tests, muscle hypertrophy, fat fraction in muscle tissue and contractility of the muscles, compared with healthy controls, will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age <18 years
* Molecularly verified MC (Thomsens or Beckers disease)

Exclusion Criteria:

* Conditions that may impair results of the study, evaluated by the investigator
* Clausphobia
* Pregnancy or breastfeeding
* Metallic objects in and around the body that are not MR-compatible

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 patients (Thomsens MC, n=20; Beckers MC, n=20) will be included along with 20 healthy age- and gender-matched controls. Inclusion criteria are age >18 years, verified MC diagnosis. Exclusion criteria areknown competing disorders that can interfere with the results (ie. muscular diseases or arthritis) or MRI contraindications.
  Before participation patients are asked about medication status. Participants who are treated for their myotonic symptoms with either Mexiletin or Lamotrigin are asked to pause their medication four days prior to participation.
  All patients will be asked to evaluate the severity of their myotonic symptoms using the MBS (Myotonic Behaviour Scale) rating from 1 (least severe) to 6 (most severe).
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Contractile properties | 1 year
  To investigate if contractile properties of the muscles are impaired in MC patients compared with healthy controls.

SECONDARY OUTCOMES:
Measuring muscle hypertrophy in upper and lower limbs | 1 year
  Visualizing and measuring hypertrophy on MRI of affected muscles in the forearm, thigh and calf of MC patients compared with muscles in healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Jacobsen, BSc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No